CLINICAL TRIAL: NCT06246461
Title: Clinical Effect Analysis of Different Regimens of Capecitabine in the Treatment of Patients With Advanced Colon Cancer
Brief Title: The Therapeutic Effect of Different Doses of Capecitabine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jingjiang People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JJPH-001
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Capecitabine
Keywords: Capecitabine; Advanced colon cancer; Clinical efficacy; Adverse reactions
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the control group: a total daily dose of 2,500 mg/m2 (Experimental): The control group was treated with capecitabine at a conventional dose: 1,250 mg/m2 orally twice daily (once in the morning and once in the evening; equivalent to a total daily dose of 2,500 mg/m2). Treatment was given for 2 weeks, followed by a 1 week of discontinuation, with each cycle lasting 3 weeks, and there were a total of 4 cycles. Administration: Swallow the tablet whole with water 30 min after breakfast and dinner every day.
  Interventions: Drug: capecitabine
- the medium-dose group: a total daily dose of 2,000 mg/m2 (Active Comparator): The medium-dose group was treated with medium-dose capecitabine: 1,000 mg/m2 orally twice daily (once in the morning and once in the evening; equivalent to a total daily dose of 2,000 mg/m2). Treatment was given for 2 weeks, followed by a 1 week of discontinuation, with each cycle lasting 3 weeks, and there were a total of 4 cycles. Administration: Swallow the tablet whole with water 30 min after breakfast and dinner every day.
  Interventions: Drug: capecitabine
- the low-dose group: a total daily dose of 1,500 mg/m2 (Active Comparator): The low-dose group was treated with low-dose capecitabine: 750 mg/m2 orally twice daily (once in the morning and once in the evening; equivalent to a total daily dose of 1,500 mg/m2). Treatment was given for 3 weeks per cycle, with each cycle lasting 3 weeks, and there were a total of 4 cycles. Administration: Swallow the tablet whole with water 30 min after breakfast and dinner every day.
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: capecitabine — The control group was treated with 2,500 mg/m2 capecitabine, with 2,000 mg/m2 capecitabine for the medium-dose group and 1,500 mg/m2 capecitabine for the low-dose group.

SUMMARY:
To observe the clinical efficacy and adverse reactions of capecitabine in the treatment of advanced colon cancer. A total of 150 patients with advanced colon cancer were selected by convenience sampling and then were divided into the control group (n = 50), the medium-dose group (n = 50), and the low-dose group (n = 50) using a random number table.Different administration regimens of capecitabine were given, and the treatment course was appropriately extended. The therapeutic effect and incidence of adverse reactions were observed.

DETAILED DESCRIPTION:
To observe the clinical efficacy and adverse reactions of capecitabine in the treatment of advanced colon cancer. A total of 150 patients with advanced colon cancer were selected by convenience sampling and then were divided into the control group (n = 50), the medium-dose group (n = 50), and the low-dose group (n = 50) using a random number table.The control group was treated with 2,500 mg/m2 capecitabine, with 2,000 mg/m2 capecitabine for the medium-dose group and 1,500 mg/m2 capecitabine for the low-dose group. Afterward, the response rate, quality of life, and adverse reactions of the three groups were collected for comparison.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria for colon cancer in the Consensus on Screening, Diagnosis and Treatment of Early Colorectal Cancer and Precancerous Lesions in China , colon cancer was confirmed by pathology
* TNM(tumor node metastasis) clinical stage was III or IV
* Predicted survival period > 3 months

Exclusion Criteria:

* Patients with heart, liver, kidney and other important organ failure and contraindications to chemotherapy
* Patients who received other anti-tumor therapy before admission
* The disease progressed rapidly and could not be successfully completed by this researcher
* Allergic to related drugs

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy:Overall response rate(RR%) | After the end of all treatment cycles (3 weeks per cycle, a total of four cycles, totaling 84 days)
  Overall response rate (RR%): complete response (CR) + partial response (PR)/total number of cases×100%.
Clinical efficacy:Disease control rate(DR)% | After the end of all treatment cycles (3 weeks per cycle, a total of four cycles, totaling 84 days)
  Disease control rate (DR)% = (CR+PR+SD)/total number of cases×100%.
Quality of life：QLQ-C30(Quality of Life Questionnaire-core30) Score | After the end of all treatment cycles (3 weeks per cycle, a total of four cycles, totaling 84 days)
  Quality of life was scored using the QLQ-C30 (Quality of Life Questionnaire-core30).QLQ-C30 is composed of one global quality of life scale and five functional scales, which include physical function, role function, emotional function, cognitive function, and social function. Scoring criteria: After the scores of each part of the scale were converted to standardized scores, the scores ranged from 0 to 100, and the higher the score of the scale, the better the overall quality of life and functional status.
Incidence of adverse reactions | After the end of all treatment cycles (3 weeks per cycle, a total of four cycles, totaling 84 days)
  Adverse reactions include hand-foot syndrome, stomatitis, leukopenia, nausea and vomiting, bone marrow suppression, and pigmentation. Incidence of adverse reactions%=number of adverse reaction cases/total number of cases × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical effect analysis of different regimens of capecitabine in the treatment of patients with advanced colon cancer, Jingjiang, Jiangsu, China

REFERENCES:
- [Derived] Ju F, Chen K, Yin D. Clinical effect analysis of different regimens of capecitabine in the treatment of patients with advanced colon cancer. J Chemother. 2025 Sep;37(5):426-435. doi: 10.1080/1120009X.2024.2385254. Epub 2024 Aug 12. PMID 39132982